CLINICAL TRIAL: NCT05184179
Title: A Multi-center, Prospective, Observational Study to Evaluate the Therapeutic Effectiveness and Safety of Olomax Tab. for Patients With Hypertension and Dyslipidemia
Brief Title: Observational Study to Evaluate the Therapeutic Effectiveness and Safety of Olomax Tab
Status: Completed | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DWJ1351_P402
Record Dates: First submitted 2021-09-03; First posted 2022-01-11 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Hypertension; Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias | interventions — Olmesartan Medoxomil

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Olmesartan Medoxomil — Olmesartan Medoxomil, Amoldipine Besylate, Rosuvastatin Ca
  Other Names: Amoldipine Besylate; Rosuvastatin Ca

SUMMARY:
Throughout this study, the efficacy and safety information of Olomax tablets will be collected from 24 weeks to 48 weeks(+8 weeks) The Data collection point is baseline, at more than 24 weeks, at more than 48 weeks(+8 weeks).

DETAILED DESCRIPTION:
The study will start after investigator determines the administration of Olomax tablets based on the investigator's judgement and obtaining informed consent from the subject during subject's daily visit.

The dose of the Olomax tablet for each subject will be determined based on efficacy and drug resistance according to the subject's previous drug administration.

Throughout this study, the efficacy and safety information of Olomax tablets will be collected from 24 weeks to 48 weeks(+8 weeks) The Data collection point is baseline, at more than 24 weeks, at more than 48 weeks(+8 weeks).

Efficacy of Olomax tablets will be evaluated based on the data collected from more than 24 weeks to 48 weeks(+8 weeks) from the baseline visit. Safety of Olomax tablets will be evaluated based on the adverse events collected during the study peroid.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over the age of 19
2. Patients eligible for Olomax Tab. prescription in accordance with the approved product manual in Korea
3. Patients who are determined to prescribe Olomax Tab. at the discretion of the investigators.

   * Antihypertensive agent: Do not include more than 3 agents.
   * Anti-abnormal lipidemia: Do not include more than 2 agents.
   * Subjects who are already administered beta blocker (BB) or diuretics due to other diseases such as angina, not for the purpose of treating hypertension may be included.
4. Consent on the use of information by the patient

Exclusion Criteria:

1. Patients who have already administered olomax tablets.
2. Subject who fall under ' Do not administer to the following patients' in the precautions for use
3. A patient who does not meet the inclusion/exclusion criteria participates
4. The patient withdraws consent for the study
5. The administration of the study drug is discontinued
6. It is impossible to follow up during the observation period
7. The investigator determines that it is no longer feasible to continue the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The number of patients was calculated based on the analysis results of the blood pressure treatment goal achievement rate and LDL-C treatment goal acheivement rate in the Olomax Tertiary Clinical Trial.
  n=(〖Z_(α/2)〗^2×p(1-p))/d^2
  :: Type 1 error (=0.05) p: Target Reach Rate at 24+ Weeks (=80%) d: Sampling error
  herefore, it means that the total number of patients required to be 95% confident that the proportion of patients whose two primary evaluation variables, blood pressure and LDL, will be included in 79-81%. Considering the dropout rate of about 20%, a total of 7,684 patients are required, so in this study, approximately 8,000 patients approximating this are finally recruited.
Sampling Method: Non-Probability Sample
Enrollment: 5450 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
Blood pressure treatment goal achievement rate | more than 24 weeks
  Blood pressure treatment goal achievement rate: The percentage of patients observed for more than 24 weeks compared to the baseline whose blood pressure reached the target value
LDL-C treatment goal achievement rate | more than 24 weeks
  LDL-C treatment goal achievement rate: The percentage of patients observed for more than 24 weeks compared to the baseline whose LDL-C reached the target level

SECONDARY OUTCOMES:
Change in blood pressure | 24 to 48 weeks
  Change in blood pressure at 24 to 48 weeks compared to baseline
The proportion of patients who have reached the treatment goal at baseline and maintain the change in blood pressure and treatment goal | 24 to 48 weeks
  The proportion of patients who have reached the treatment goal at baseline and maintain the change in blood pressure and treatment goal at 24 to 48 weeks
the percentage of patients maintaining the treatment goal and the amount of change in blood pressure | 24 to 48 weeks
  Among patients who reached the treatment goal at baseline, the percentage of patients maintaining the treatment goal and the amount of change in blood pressure at 24 to 48 weeks for each antihypertensive drug (single, double drug combination classification)
Patients who did not reach the treatment goal at baseline, change in blood pressure and rate of reaching the treatment goal | 24 to 48 weeks
  Patients who did not reach the treatment goal at baseline, change in blood pressure and rate of reaching the treatment goal at 24 to 48 weeks
For patients who did not reach the treatment goal at baseline, the amount of change in blood pressure and the rate of reaching the treatment goal | 24 to 48 weeks
  For patients who did not reach the treatment goal at baseline, the amount of change in blood pressure and the rate of reaching the treatment goal at 24 to 48 weeks by antihypertensive drug (single, combined classification)
Change in LDL-C | 24 to 48 weeks
  Change in LDL-C at 24 to 48 weeks compared to baseline
Among patients who reached the treatment goal at baseline, the change in LDL-C, the proportion of patients maintaining the treatment goal | 24 to 48 weeks
  Among patients who reached the treatment goal at baseline, the change in LDL-C at 24 to 48 weeks and the proportion of patients maintaining the treatment goal
Among patients who reached the treatment goal at baseline, the change in LDL-C , the proportion of eligible patients maintaining the treatment goal | 24 to 48 weeks
  Among patients who reached the treatment goal at baseline, the change in LDL-C at 24 to 48 weeks for each anti-dyslipidemia agent and the proportion of eligible patients maintaining the treatment goal
For patients who did not reach the treatment goal at baseline, change in LDL-C, rate of reaching the treatment goal | 24 to 48 weeks
  For patients who did not reach the treatment goal at baseline, change in LDL-C and rate of reaching the treatment goal at 24 to 48 weeks
For patients who did not reach the treatment goal at baseline, change in LDL-C, rate of reaching the treatment goal | 24 to 48 weeks
  For patients who did not reach the treatment goal at baseline, change in LDL-C and rate of reaching the treatment goal at 24 to 48 weeks for each anti-dyslipidemia agent
Change amount and rate of change in lipid variables | 24 to 48 weeks
  Change amount and rate of change in lipid variables (Non-HDL, HDL-C, TG, TC) at 24 to 48 weeks compared to the baseline
the rate and amount of change in both blood pressure and LDL-C | more than 24 weeks
  Patients who underwent FU for more than 24 weeks compared to the baseline, the rate and amount of change in both blood pressure and LDL-C reached the target values
Change in Framingham Risk Score (FRS) | more than 24 weeks
  Change in Framingham Risk Score (FRS) over 24 weeks compared to baseline
change in carotid intima-media thickening (CIMT) value | more than 24 weeks
  If data exists, change in carotid intima-media thickening (CIMT) value over 24 weeks compared to baseline
hsCRP change | more than 24 weeks
  If information is collected, hsCRP change over 24 weeks compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Undecided